CLINICAL TRIAL: NCT03985774
Title: The ENROUTE Transcarotid Neuroprotection System (ENROUTE Transcarotid NPS) DW-MRI Study
Acronym: DW-MRI OUS
Status: Completed | Type: Observational
Sponsor: Silk Road Medical (Industry)
Collaborators: Complejo Hospitalario Toledo (Other); University Ghent (Other); Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: SRM-2014-03
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Carotid Stenosis; Carotid Artery Diseases; Carotid Atherosclerosis; Carotid Artery Plaque
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients requiring carotid revascularization: Symptomatic patients, male or female, with atherosclerotic extracranial internal carotid stenosis (ICA) with or without involvement of the contiguous common artery (CCA), that require carotid revascularization.
  Interventions: Procedure: Transcarotid revascularization

INTERVENTIONS:
Procedure: Transcarotid revascularization — The ENROUTE Transcarotid Neuroprotection System (NPS) has received CE Mark and is commercially available in the European Union. The ENROUTE Transcarotid NPS may be used in conjunction with carotid artery stent approved for revascularization in patients with carotid disease The ENROUTE Transcarotid Neuroprotection System is intended to provide transcarotid vascular access, introduction of diagnostic agents and therapeutic devices, and embolic protection during carotid artery angioplasty and stenting procedures for patients diagnosed with carotid artery stenosis
  Other Names: Transcarotid Revascularization (TCAR); Carotid Artery Stenting

SUMMARY:
The goal of this study is to evaluate the incidence of post procedure DW-MRI lesions (relative to baseline) and debris captured in the ENROUTE Transcarotid NPS inline filter during a transcarotid stenting procedure.

DETAILED DESCRIPTION:
The ENROUTE Transcarotid NPS has received CE Mark and is commercially available in the European Union. The ENROUTE Transcarotid NPS may be used in conjunction with carotid artery stent approved for revascularization in patients with carotid disease in the context of this study.

This is a prospective, single-arm, multi-center clinical trial of the ENROUTE Transcarotid NPS in conjunction with all commercially approved carotid artery stents used for revascularization in patients with carotid disease.

The goal of this study is to evaluate the incidence of post procedure DW-MRI lesions (relative to baseline) and debris captured in the ENROUTE Transcarotid NPS inline filter during a transcarotid stenting procedure.

A patient is considered enrolled after:

1. meeting all inclusion and none of the exclusion criteria,
2. the transcarotid arterial sheath has entered into the patient's vasculature. Insertion of the venous sheath does not qualify a patient as enrolled.

Patients who are screened but do not meet all study criteria are considered screen failures and may not be enrolled. Patients in whom an arterial sheath is placed but who do not meet all study entry criteria are considered enrolled.

The Investigator is responsible for maintaining any information pertaining to the Ethics Committee review and approval as required by local law.

ELIGIBILITY:
Inclusion Criteria:

* Patient is symptomatic and has a history of stroke (minor or non-disabling), TIA and/or amaurosis fugax within 60 days of the procedure.
* Target vessel must meet diameter requirements for stent (refer to selected stent IFU for diameter requirements).
* Patient has a discrete lesion located in the internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA).
* Patient is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.

Exclusion Criteria:

* Patient has chronic atrial fibrillation.
* Patient has had any episode of paroxysmal atrial fibrillation within the past 6 months, or history of paroxysmal atrial fibrillation requiring chronic anticoagulation.
* Patient has an evolving stroke.
* Patient has a history of spontaneous intracranial hemorrhage within the past 12 months.
* Patient has had a recent (<7 days) stroke of sufficient size (on CT or MRI) to place him or her at risk of hemorrhagic conversion during the procedure.
* Patient had hemorrhagic transformation of an ischemic stroke within the past 60 days.
* Patient has active bleeding diathesis or coagulopathy or will refuse blood transfusion.
* Patient had or will have CABG, endovascular stent procedure, valve intervention or vascular surgery within 30 days before or after the intervention.
* Patient has had a recent GI bleed that would interfere with antiplatelet therapy.
* Patient has history of intolerance or allergic reaction to any of the study medications or stent materials (refer to stent IFU), including aspirin (ASA), ticlopidine, clopidogrel, prasugrel, statin or contrast media (that can't be pre medicated). Patients must be able to tolerate statins and a combination of ASA and ticlopidine, ASA and clopidogrel or ASA and prasugrel.
* Patient with a history of major stroke (CVA) with major neurological deficit likely to confound study endpoints within 1 month of index procedure.
* Patient has an intracranial tumor.
* Patient is actively participating in another drug or device trial (IND or IDE) that has not completed the required protocol follow-up period.
* Patient has inability to understand and cooperate with study procedures.
* Occlusion or [Thrombolysis In Myocardial Infarction Trial (TIMI 0)] "string sign" >1cm of the ipsilateral common or internal carotid artery.
* Confirmed and uncorrected cardiac sources of emboli.
* Patient has a prosthetic heart valve
* Ostium of Common Carotid Artery (CCA) requires revascularization.
* Presence of extensive or diffuse atherosclerotic disease involving the proximal common carotid artery that would preclude the safe introduction of the study device.
* The patient has less than 5cm between the clavicle and bifurcation, as assessed by duplex Doppler ultrasound.
* Bilateral carotid stenosis if intervention is planned within 37 days of the index procedure.
* An intraluminal filling defect (defined as an endoluminal lucency surrounded by contrast, seen in multiple angiographic projections, in the absence of angiographic evidence of calcification) that is not associated with an ulcerated target lesion.
* Abnormal angiographic findings: ipsilateral intracranial or extracranial arterial stenosis greater in severity than the lesion to be treated, cerebral aneurysm > 5 mm, AVM (arteriovenous malformation) of the cerebral vasculature, or other abnormal angiographic findings.
* Patient has had a previous intervention in the ipsilateral proximal CCA.
* Patient is otherwise unsuitable for intervention in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled into this study will be comprised of male and female symptomatic patients requiring carotid revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
New White Lesions | 30 days
  Incidence of new white lesions by DW-MRI post procedure.

SECONDARY OUTCOMES:
Periprocedural SAEs | 30 days
  All stroke
Periprocedural SAEs | 30 days
  All death
post-procedure filter debris | 30 days
  filter debris morphology
DW-MRI Lesions | 30 days
  Location of DW-MRI lesions
DW-MRI Lesions | 30 days
  Volume of DW-MRI lesions

CONTACTS AND LOCATIONS:
Locations (3):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Technischen Universitat Munchen, Munich, Germany
- Complejo Hospitalario de Toledo, Toledo, Spain